CLINICAL TRIAL: NCT01156701
Title: Prophylactic Efficacy of Relenza Against Influenza A and B
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113502; WEUSRTP2058; EPI40499
Record Dates: First submitted 2010-04-22; First posted 2010-07-05 (Estimated); Results first posted 2011-03-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bronchospasm; Influenza, Human; Asthma; Respiratory Disease; Exacerbation of COPD; Bronchitis; Otitis Maedia; Pneumonia; Sinusitis
Keywords: Influenza; Zanamivir; Influenza prophylaxis; Relenza
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchial Spasm; Influenza, Human; Asthma; Respiration Disorders; Bronchitis; Pneumonia; Sinusitis | interventions — Zanamivir

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort1: Prophylaxis with untreated index: Individuals are eligible to be included in the prophylaxis with untreated index cohort if they are at least 5 years old and have at least 6 months of continuous enrollment, and
  1. Received a dispensing of Relenza (HICL=020398 or HCPCS = G9018 or G9034), and
  2. Have no diagnosis of influenza (ICD-9 487.xx) on the day of Relenza dispensing or in the 3 preceding days, and
  3. A household member (index case) with the same family identifier code has had a medical visit (outpatient, inpatient or emergency room (ER) visit) in the 3 days preceding or the day of the Relenza dispensing with a diagnosis of influenza (ICD-9 487.xx), and
  4. The household member (index case) has not received any antiviral therapy (oseltamivir (Tamiflu), rimantadine, amantadine, and zanamivir (Relenza)) on the day of or the day after the index case's medical visit associated with a diagnosis of influenza.
  Interventions: Drug: Receiving a prescription of Relenza for prophylaxis
- Cohort2: Prophylaxis with treated index: Individuals are eligible to be included in the prophylaxis with treated index cohort if they are at least 5 years old, have 6 months continuous enrollment and
  1. Received a dispensing of Relenza (HICL=020398 or HCPCS = G9018 or G9034), and
  2. Have no diagnosis of influenza (ICD-9 487.xx) on the day of Relenza dispensing or in the 3 preceding days, and
  3. A household member (index case) with the same family ID variable has had a medical visit (outpatient, inpatient or ER visit) in the 3 days preceding or the day of the Relenza dispensing with a diagnosis of influenza (ICD-9 487.xx), and
  4. The household member (index case) has received any antiviral therapy (oseltamivir (Tamiflu), rimantadine, amantadine, and zanamivir (Relenza)) on the day of or the day after the index case's medical visit associated with a diagnosis of influenza.
  Interventions: Drug: Receiving a prescription of Relenza for prophylaxis
- Cohort3: No prophylaxis with untreated index: Individuals are eligible to be included in the no prophylaxis with untreated index cohort if they are at least 5 years old, have 6 months continuous enrollment and
  1. Have not received a dispensing of Relenza (HICL=020398 or HCPCS = G9018 or G9034) within 3 days following the date on which
  2. A household member (index case) with the same family ID variable has had a medical visit (outpatient, inpatient or ER visit) with a diagnosis of influenza (ICD-9 487.xx), and
  3. The household member (index case) has not received any antiviral therapy (oseltamivir (Tamiflu), rimantadine, amantadine, and zanamivir (Relenza)) on the day of or the day after the index case's medical visit associated with a diagnosis of influenza.
  Interventions: Other: No prophylaxis with Relenza
- Cohort4: No prophylaxis with treated index: Individuals are eligible to be included in the no prophylaxis with treated index cohort if they are at least 5 years old, have 6 months continuous enrollment and
  1. Have not received a dispensing of Relenza(HICL=020398 or HCPCS = G9018 or G9034) within 3 days following the date on which
  2. A household member (index case) with the same family ID variable has had a medical visit (outpatient, inpatient or ER visit) with a diagnosis of influenza (ICD-9 487.xx), and
  3. The household member (index case) has received zanamivir (Relenza) on the day of or the day after the index case's medical visit associated with a diagnosis of influenza
  Interventions: Other: No prophylaxis with Relenza

INTERVENTIONS:
Drug: Receiving a prescription of Relenza for prophylaxis — Receiving a prescription of Relenza for prophylaxis
  Groups: Cohort1: Prophylaxis with untreated index; Cohort2: Prophylaxis with treated index
Other: No prophylaxis with Relenza — No prophylaxis with Relenza
  Groups: Cohort3: No prophylaxis with untreated index; Cohort4: No prophylaxis with treated index

SUMMARY:
In response to the European regulatory authorities, GSK is conducting a post-marketing observational study to assess the efficacy of Relenza when used as prophylaxis against influenza.

SPECIFIC AIMS

1. Determine the frequency of patients who received Relenza from October 2006 through April 2009, and among them the number who have no concurrent diagnosis of influenza, i.e., those receiving Relenza for prophylaxis, and among these the number who have a family member with a medical visit for influenza within three days preceding the above indentified patient's dispensing of Relenza. This is to determine the feasibility of conducting detailed analysis.
2. If analysis is feasible then tabulate the frequency of influenza-like-illness and respiratory outcomes in users of prophylactic Relenza and their family members and in family members of persons using Relenza for the treatment of influenza (i.e., index cases).
3. If analysis is feasible then estimate the direct effect of prophylactic Relenza on the occurrence of influenza-like-illness and respiratory outcomes, the secondary effect of Relenza treatment of influenza on susceptible family members, and the total effect of Relenza (treatment plus prophylaxis).

METHODS Overview of Study Design This is an analysis of the 30-day risk of influenza-like illness and respiratory outcomes in persons for whom some household members (index cases) have had a medical visit associated with a diagnosis of influenza. The exposed individuals to the index case will be categorized into one of four cohorts according to whether the exposed person received prophylactic Relenza or no antiviral treatment and by whether the index family member with a diagnosis of influenza received antiviral treatment.

Estimates of the direct effect of Relenza prophylaxis, the indirect effectof preventing disease in susceptible family members, and the total effect of disease reduction when both index cases and susceptible family members are treated will be obtained from different comparisons between cohorts, as outlined below.

The research will cover the first three influenza seasons during which Relenza has been indicated for prophylactic use in the United States. These will be from October through April of 2006-2009.

DETAILED DESCRIPTION:
***Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.***

This analysis will use the i3 Ingenix proprietary National Health Information (NHI) database, containing claims and enrollment data back to 1993, with the opportunity to link patient and physician survey data to pharmacy and medical claims, and clinical laboratory results. These data are use for a wide range of pharmacoepidemiologic, healthcare utilization, and economic analyses. In addition to data derived from affiliated health plans, data from large, national employer groups are also stored in the database. The data undergo regular audits and quality control procedures. The accessible information includes demographics, pharmacy use, and all medical and facilities claims, which provide data on services, procedures, and their accompanying diagnoses. Underlying information is geographically diverse across the US, and is updated frequently. The insured population from which the database draws the data comprises approximately 4 percent of the US population. The data used for analysis is de-identified.

Study Cohorts From October 2006 through April 2009, we will count patients receiving prophylactic Relenza, defined as a dispensing of Relenza to a person who meets two criteria: (1) not having had a diagnosis of influenza associated with medical care on the day of dispensing or in the preceding three days, and (2) a household member has had a diagnosis of influenza associated with medical care on the day of the index dispensing or within the preceding three days. "Household members" will be defined operationally as persons within the RDM sharing a common family identifier and address.

We will assemble the study cohorts for the 3 influenza seasons running from October 2006 through April 2009. Cohort membership is based on the treatment an individual receives and the nature of household exposure.

Exclusion criteria include:

* Sex unknown
* Year of birth is missing or where the date of dispensing or service date preceded the year of birth
* Age at index date is less than 5 years
* Not enrolled in the health plan for 6 months prior to the study entry date

Observation begins for the prophylaxis and treated patients on the day following Relenza dispensing and for the non-prophylaxis and untreated patients on the third day following their medical visit, and continues for a total of 30 days.

Covariates For each individual we will identify age, sex, medical conditions requiring care in the six months preceding cohort entry from insurance claims for health services. Medical conditions requiring care will be defined at the 3-digit ICD9 diagnostic level.

Outcomes We will identify medical visits and hospitalizations with influenza-like illness and respiratory disease in the 30 days following cohort entry.

Analysis

Within categories of age of 5-14, 15-44, 45-64 and 65+ years, we will tabulate:

* the number of individuals in each of four cohorts (cohorts defined below)
* the number of medical visits for influenza-like illness and respiratory illness in the 30-day follow-up period

For each outcome we will estimate the following antiviral efficacy measures detailed in Halloran's analysis of clinical trials data [Halloran, 2007]. The first two effects below will be standardization to the age distribution of all persons receiving prophylactic Relenza;

1. Direct Effect of Relenza Prophylaxis: Risk in Cohort 1 is less than Risk in Cohort 3 Prophylaxis patient with untreated index case vs patient without prophylaxis with untreated index
2. Total Effect of Relenza Prophylaxis and Treatment: Risk in Cohort 2 is less than Risk in Cohort 3 Prophylaxis patient with treated index case vs. patient without prophylaxis with untreated index

   We will calculate the following effect estimate with standardization to the age distribution of untreated persons.
3. Protective Effect of Relenza Prophylaxis on Susceptible: Risk in Cohort 2 is less than Risk in Cohort 4 Prophylaxis patient with treated index case vs. patient without prophylaxis with treated index

Using binomial regression and a linear risk model, we will obtain adjusted estimates for Direct Effect, Total Effect, and Protective Effect, defined as above, adjusted for age group, sex, and any diagnosis with a prevalence of at least 10 percent in the cohorts combined.

ELIGIBILITY:
Inclusion Criteria:

* 5 years or older
* At least 6 months of continuous follow up time
* Received Relenza without a diagnosis of influenza

Exclusion Criteria:

* Sex unknown
* Year of birth is missing
* Date of dispensing or service date preceded the year of birth
* Age at index date is less than 5 years
* Not enrolled in the health plan for 6 months prior to the study entry date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will use data from the NHI database which includes only those individuals who have both medical and pharmacy benefits, and therefore captures most outpatient prescription drug exposures and health provider encounters. From October 2006 through April 2009, we will count patients receiving prophylactic Relenza, defined as a dispensing of Relenza to a person who meets 2 criteria: (1) not having had a diagnosis of influenza associated with medical care on the day of dispensing or in the preceding 3 days, and (2) a household member has had a diagnosis of influenza associated with medical care on the day of the prophylactic dispensing or within the preceding 3 days. Household members will be defined as persons within the NHI database sharing a common family identifier code.
Sampling Method: Non-Probability Sample
Enrollment: 171705 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Result] Kandace Amend, Vani Vannappagari, Maria Wood-Armany, Rob Gately, John Seeger; Effectiveness of Zanamivir Prophylaxis for Influenza.26th ICPE: International Conference on Pharmacoepidemiology & Therapeutic Risk Management August 19-22, 2010, Brighton, UK

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Prophylaxis With Untreated Index: Individuals who received zanamivir prophylaxis and who had a household member who had a medical visit with a diagnosis of influenza and did not receive antiviral therapy (oseltamivir, rimantidine, amantidine, or zanamivir)
- Cohort 2: Prophylaxis With Treated Index: Individuals who received zanamivir prophylaxis and who had a household member who had a medical visit with a diagnosis of influenza and received antiviral therapy (oseltamivir, rimantidine, amantidine, or zanamivir)
- Cohort 3: Untreated With Untreated Index: Individuals not receiving zanamivir prophylaxis and who had a household member who had a medical visit with a diagnosis of influenza and did not receive any antiviral therapy (oseltamivir, rimantidine, amantidine, or zanamivir)
- Cohort 4: Untreated With Treated Index: Individuals not receiving zanamivir prophylaxis and who had a household member who had a medical visit with a diagnosis of influenza and received zanamivir on the day of or the day after the influenza diagnosis
Period: Overall Study
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Started | 257 | 1007 | 163716 | 6725
Completed | 257 | 1007 | 163716 | 6725
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients Included in the Analysis: All patients at least 5 years old enrolled for at least 6 months in the Normative Health Informatics (NHI) insurance claims database during the influenza seasons of 2006-2009
Arm/Group | All Patients Included in the Analysis
Number analyzed (Participants) | 171705
Age, Customized [Number; unit: Participants] — Number of participants in the indicated age category
  Participants
    5-14 years | 47670
    15-44 years | 85640
    45-64 years | 37119
    >=65 years | 1276
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84162
  Male | 87543

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Influenza
Description: The frequency of influenza among the four cohorts was measured.
Time Frame: 2006-2009
Population: The study population consisted of individuals who were at least 5 years old and had been continuously enrolled for at least 6 months in the Normative Health Informatics (NHI) insurance claims database during the influenza seasons of 2006-2009 (October-April).
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Influenza | 3 | 10 | 2539 | 93
  No Influenza | 254 | 997 | 161177 | 6632
Statistical Analysis 1: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.15, 95% CI 2-sided [-1.42 to 1.12] — Direct effect of Zanamivir prophylaxis on influenza risk
Statistical Analysis 2: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.38, 95% CI 2-sided [-0.93 to 0.17] — Total effect of zanamivir prophylaxis
Statistical Analysis 3: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.14, 95% CI 2-sided [-0.75 to 0.47] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 4: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = 0.23, 95% CI 2-sided [-1.15 to 1.62] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 5: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.24, 95% CI 2-sided [-0.51 to 0.03] — Protective effect of zanamivir on susceptible risk
Statistical Analysis 6: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.01] — Direct effect of Zanamivir prophylaxis on influenza risk
Statistical Analysis 7: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Total effect of zanamivir prophylaxis
Statistical Analysis 8: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 9: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.02] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 10: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Protective effect of zanamivir on susceptible risk

2. Secondary Outcome: Number of Patients With Asthma
Description: The frequency of asthma among the four cohorts was measured.
Time Frame: 2006-2009
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Asthma | 1 | 5 | 1488 | 54
  No Asthma | 256 | 1002 | 162228 | 6671
Statistical Analysis 1: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.40, 95% CI 2-sided [-1.17 to 0.36] — Direct effect of Zanamivir prophylaxis on asthma risk
Statistical Analysis 2: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.38, 95% CI 2-sided [-0.80 to 0.03] — Total effect of zanamivir prophylaxis
Statistical Analysis 3: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.28, 95% CI 2-sided [-0.75 to 0.18] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 4: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.02, 95% CI 2-sided [-0.89 to 0.85] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 5: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.10, 95% CI 2-sided [-0.31 to 0.11] — Protective effect of zanamivir on susceptible risk
Statistical Analysis 6: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Direct effect of Zanamivir prophylaxis on asthma risk
Statistical Analysis 7: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Total effect of zanamivir prophylaxis
Statistical Analysis 8: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 9: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.01] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 10: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [1.00 to 1.00] — Protective effect of zanamivir on susceptible risk

3. Secondary Outcome: Number of Patients With Pneumonia
Description: The frequency of pneumonia among the four cohorts was measured..
Time Frame: 2006-2009
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Pneumonia | 2 | 1 | 541 | 16
  No Pneumonia | 255 | 1006 | 163175 | 6709
Statistical Analysis 1: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = 0.46, 95% CI 2-sided [-0.61 to 1.54] — Direct effect of Zanamivir prophylaxis on pneumonia risk
Statistical Analysis 2: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.45 to -0.04] — Total effect of zanamivir prophylaxis
Statistical Analysis 3: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.15, 95% CI 2-sided [-0.39 to 0.09] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 4: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = 0.72, 95% CI 2-sided [-0.38 to 1.81] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 5: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.10, 95% CI 2-sided [-0.22 to 0.02] — Protective effect of zanamivir on susceptible risk
Statistical Analysis 6: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.02] — Direct effect of Zanamivir prophylaxis on pneumonia risk
Statistical Analysis 7: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [1.00 to 1.00] — Total effect of zanamivir prophylaxis
Statistical Analysis 8: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [1.00 to 1.00] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 9: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.01, 95% CI 2-sided [1.00 to 1.02] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 10: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [1.00 to 1.00] — Protective effect of zanamivir on susceptible risk

4. Secondary Outcome: Number of Patients With Bronchitis
Description: The frequency of bronchitis among the four cohorts was measured.
Time Frame: 2006-2009
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Bronchitis | 8 | 15 | 2572 | 96
  No Bronchitis | 249 | 992 | 161144 | 6629
Statistical Analysis 1: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = 1.28, 95% CI 2-sided [-0.83 to 3.40] — Direct effect of Zanamivir prophylaxis on bronchitis risk
Statistical Analysis 2: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.24, 95% CI 2-sided [-0.98 to 0.47] — Total effect of zanamivir prophylaxis
Statistical Analysis 3: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.09, 95% CI 2-sided [-0.85 to 0.67] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 4: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = 1.53, 95% CI 2-sided [-0.70 to 3.76] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 5: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.16, 95% CI 2-sided [-0.44 to 0.12] — Protective effect of zanamivir on susceptible risk
Statistical Analysis 6: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.99 to 1.03] — Direct effect of Zanamivir prophylaxis on bronchitis risk
Statistical Analysis 7: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Total effect of zanamivir prophylaxis
Statistical Analysis 8: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.01] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 9: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.99 to 1.04] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 10: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [1.00 to 1.00] — Protective effect of zanamivir on susceptible risk

5. Secondary Outcome: Number of Patients With Any Respiratory Diagnosis
Description: The frequency of any respiratory diagnosis among the four cohorts was measured.
Time Frame: 2006-2009
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Respiratory Diagnosis | 16 | 50 | 10166 | 420
  No Respiratory Diagnosis | 241 | 957 | 153550 | 6305
Statistical Analysis 1: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.14, 95% CI 2-sided [-3.08 to 2.79] — Direct effect of Zanamivir prophylaxis on risk of any respiratory diagnosis
Statistical Analysis 2: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Difference (RD) = -1.07, 95% CI 2-sided [-2.39 to 0.25] — Total effect of zanamivir prophylaxis
Statistical Analysis 3: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -1.08, 95% CI 2-sided [-2.51 to 0.35] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 4: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = 0.93, 95% CI 2-sided [-2.29 to 4.14] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 5: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.58 to 0.59] — Protective effect of zanamivir on susceptible risk
Statistical Analysis 6: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.97 to 1.03] — Direct effect of Zanamivir prophylaxis on risk of any respiratory diagnosis
Statistical Analysis 7: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 3: Untreated With Untreated Index; Test type: Superiority or Other; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.98 to 1.00] — Total effect of zanamivir prophylaxis
Statistical Analysis 8: Comparison: Cohort 2: Prophylaxis With Treated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.98 to 1.00] — Direct effect of zanamivir prophylaxis when index is treated
Statistical Analysis 9: Comparison: Cohort 1: Prophylaxis With Untreated Index vs Cohort 2: Prophylaxis With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.98 to 1.04] — Risk in cohort 1 minus risk in cohort 2
Statistical Analysis 10: Comparison: Cohort 3: Untreated With Untreated Index vs Cohort 4: Untreated With Treated Index; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.00] — Protective effect of zanamivir on susceptible risk

6. Other Pre Specified Outcome: Number of Patients With Respiratory Outcomes
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Influenza | 3 | 10 | 2539 | 93
  Asthma | 1 | 5 | 1488 | 54
  Chronic obstructive pulmonary disease (COPD) | 0 | 0 | 153 | 3
  Exacerbation of COPD | 0 | 0 | 34 | 0
  Bronchospasm | 0 | 0 | 110 | 5
  Pneumonia | 2 | 1 | 541 | 16
  Bronchitis | 8 | 15 | 2572 | 96
  Sinusitis | 1 | 20 | 2708 | 140
  Otitis media | 2 | 4 | 1582 | 64
  Any of the above | 16 | 50 | 10166 | 420

7. Other Pre Specified Outcome: Number of Participants Experiencing Hospitalization or Death Due to Influenza
Description: The frequency of hospitalization and death in the study population was analyzed.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Number analyzed (Participants) | 257 | 1007 | 16371 | 6725
patients
  Hospitalization | 0 | 6 | 1063 | 41
  Death | 0 | 0 | 4 | 0

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Cohort 1: Prophylaxis With Untreated Index | Cohort 2: Prophylaxis With Treated Index | Cohort 3: Untreated With Untreated Index | Cohort 4: Untreated With Treated Index
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.